CLINICAL TRIAL: NCT01948518
Title: The Effect of Sildenafil on Diffusion Capacity Measurements in Patients With Pulmonary Hypertension and Parenchymal Lung Disease
Brief Title: Effect of Sildenafil on Diffusion Capacity in Patients With PH and Parenchymal Lung Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Umur Hatipoglu, MD, Staff Pulmonary, Allergy and Critical Care Medicine, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08-993
Record Dates: First submitted 2013-09-18; First posted 2013-09-23 (Estimated); Results first posted 2014-09-30 (Estimated); Last update posted 2014-09-30 (Estimated); Status verified 2014-07

CONDITIONS: Diffuse Parenchymal Lung Disease; Pulmonary Hypertension
Keywords: Pulmonary hypertension; Parenchymal Lung Disease; Diffusion Capacity
MeSH Terms: conditions — Lung Diseases, Interstitial; Hypertension, Pulmonary | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral sildenafil 20 mg (Experimental): oral sildenafil, single dose at baseline
  Interventions: Drug: Oral sildenafil 20 mg

INTERVENTIONS:
Drug: Oral sildenafil 20 mg — A single dose of sildenafil will be given after recording baseline diffusion capacity and 6 minute walk. Measurements will be repeated one hour after the drug.
  Other Names: sildenafil

SUMMARY:
The purpose of this study was to investigate the acute effects of sildenafil on diffusion capacity, a commonly performed pulmonary function test, which is used to assess the lungs' gas exchange capability.

This study does not assess safety or efficacy of the drug. The study does not have clinical end points. The variables studied are diffusion capacity and 6 minute walk after a single dose of sildenafil.

This study has been completed.

DETAILED DESCRIPTION:
Sildenafil is a cyclic GMP selective phosphodiesterase type 5 inhibitor approved for use by the FDA in patients with pulmonary arterial hypertension. There has been recent interest in the use of the drug in patients with diffuse parenchymal lung diseases. This is largely based on sildenafil's salutary effects observed in small studies (Collard et al. 897-99;Ghofrani et al. 895-900;Collard et al. 897-99) and the frequent coexistence of pulmonary hypertension in these patients (Nathan et al. 657-63). In eight patients with pulmonary fibrosis and pulmonary hypertension, sildenafil reduced pulmonary artery pressure and improved shunt fraction as determined by multiple inert gas elimination technique (Ghofrani et al. 895-900;Nathan et al. 657-63). Collard et al demonstrated a 49 meter improvement in 6 minute walk distance in 11 patients with idiopathic pulmonary fibrosis and pulmonary hypertension after 3 months of therapy with sildenafil.

Main theoretical concern with the use of pulmonary arterial vasodilator therapy has been worsening of ventilation perfusion matching due to release of hypoxic vasoconstriction. Such a phenomenon is well recognized during prostacyclin infusion(Ghofrani et al. 895-900;Walmrath et al. 1084-92). Inhaled route seems to circumvent this side effect by preferentially delivering the drug to the alveoli with high V/Q ratios and augmenting blood flow to these regions (Ghofrani et al. 895-900;Walmrath et al. 1084-92). In the only study to address possible effect of systemically administered sildenafil on gas exchange, Ghofrani et al observed improvement in V/Q matching in eight patients using the multiple inert gas elimination technique (MIGET). The authors postulated an enhancement of local defense mechanisms against hypoxia i.e. increased nitric oxide availability to hypoxic alveoli despite oral route of administration(Ghofrani et al. 895-900). In a recent study of 14 normal subjects, oral sildenafil did not effect DLCO measurements at rest, after exercise and under hypoxic conditions(Snyder et al. 421-30).

Diffusion capacity of the lung for carbon monoxide (DLCO) is the clinically available method of assessing gas exchange for practitioners. It is frequently used as a tool for serial monitoring of diffuse parenchymal lung disease. American Thoracic Society has endorsed its use in the assessment of patients with idiopathic interstitial pneumonias(American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias . This Joint Statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS Board of Directors, June 2001 and by The ERS Executive Committee, June 2001 277-304).

The aim of our study was to delineate the effects of orally administered sildenafil on diffusion capacity (absolute value). The significance of this information was twofold. First, it would be helpful clinically to determine the contribution of a pulmonary vasodilator to the change in DLCO to separate this effect from a true clinical change. Second, sildenafil's effect on gas exchange may lead to modifications in therapy such as changes in oxygen flow delivered to patients.

This is not a study that measures clinical outcome or safety of sildenafil. A single dose was administered and effect on diffusion capacity and 6 minute walk were assessed compared to baseline. While we would caution clinicians for rare exceptions to these findings, we believe our data exclude a significant confounding effect in interpretation of diffusion capacity in patients with parenchymal lung disease who are treated for pulmonary hypertension with oral sildenafil. Whether this conclusion holds true at higher doses of sildenafil and in patients with vasodilator response may offer further venues for research.

We were asked to retrospectively register the study at the request of BMC Pulmonary Medicine Journal Editorial Office prior to publication.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients over age 18 years of age who are able to consent
* Diagnosis of diffuse parenchymal lung disease with concomitant pulmonary hypertension

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2009-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Umur Hatipoglu, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Background] Lettieri CJ, Nathan SD, Barnett SD, Ahmad S, Shorr AF. Prevalence and outcomes of pulmonary arterial hypertension in advanced idiopathic pulmonary fibrosis. Chest. 2006 Mar;129(3):746-52. doi: 10.1378/chest.129.3.746. PMID 16537877
- [Background] Hamada K, Nagai S, Tanaka S, Handa T, Shigematsu M, Nagao T, Mishima M, Kitaichi M, Izumi T. Significance of pulmonary arterial pressure and diffusion capacity of the lung as prognosticator in patients with idiopathic pulmonary fibrosis. Chest. 2007 Mar;131(3):650-656. doi: 10.1378/chest.06-1466. Epub 2007 Feb 22. PMID 17317730
- [Background] Ghofrani HA, Wiedemann R, Rose F, Schermuly RT, Olschewski H, Weissmann N, Gunther A, Walmrath D, Seeger W, Grimminger F. Sildenafil for treatment of lung fibrosis and pulmonary hypertension: a randomised controlled trial. Lancet. 2002 Sep 21;360(9337):895-900. doi: 10.1016/S0140-6736(02)11024-5. PMID 12354470
- [Background] Badesch DB, Hill NS, Burgess G, Rubin LJ, Barst RJ, Galie N, Simonneau G; SUPER Study Group. Sildenafil for pulmonary arterial hypertension associated with connective tissue disease. J Rheumatol. 2007 Dec;34(12):2417-22. Epub 2007 Nov 1. PMID 17985403
- [Background] Rubin LJ, Badesch DB, Fleming TR, Galie N, Simonneau G, Ghofrani HA, Oakes M, Layton G, Serdarevic-Pehar M, McLaughlin VV, Barst RJ; SUPER-2 Study Group. Long-term treatment with sildenafil citrate in pulmonary arterial hypertension: the SUPER-2 study. Chest. 2011 Nov;140(5):1274-1283. doi: 10.1378/chest.10-0969. Epub 2011 May 5. PMID 21546436
- [Background] Idiopathic Pulmonary Fibrosis Clinical Research Network; Zisman DA, Schwarz M, Anstrom KJ, Collard HR, Flaherty KR, Hunninghake GW. A controlled trial of sildenafil in advanced idiopathic pulmonary fibrosis. N Engl J Med. 2010 Aug 12;363(7):620-8. doi: 10.1056/NEJMoa1002110. Epub 2010 May 18. PMID 20484178
- [Background] American Thoracic Society; European Respiratory Society. American Thoracic Society/European Respiratory Society International Multidisciplinary Consensus Classification of the Idiopathic Interstitial Pneumonias. This joint statement of the American Thoracic Society (ATS), and the European Respiratory Society (ERS) was adopted by the ATS board of directors, June 2001 and by the ERS Executive Committee, June 2001. Am J Respir Crit Care Med. 2002 Jan 15;165(2):277-304. doi: 10.1164/ajrccm.165.2.ats01. No abstract available. PMID 11790668
- [Background] Miller A, Thornton JC, Warshaw R, Anderson H, Teirstein AS, Selikoff IJ. Single breath diffusing capacity in a representative sample of the population of Michigan, a large industrial state. Predicted values, lower limits of normal, and frequencies of abnormality by smoking history. Am Rev Respir Dis. 1983 Mar;127(3):270-7. doi: 10.1164/arrd.1983.127.3.270. No abstract available. PMID 6830050
- [Background] Macintyre N, Crapo RO, Viegi G, Johnson DC, van der Grinten CP, Brusasco V, Burgos F, Casaburi R, Coates A, Enright P, Gustafsson P, Hankinson J, Jensen R, McKay R, Miller MR, Navajas D, Pedersen OF, Pellegrino R, Wanger J. Standardisation of the single-breath determination of carbon monoxide uptake in the lung. Eur Respir J. 2005 Oct;26(4):720-35. doi: 10.1183/09031936.05.00034905. No abstract available. PMID 16204605
- [Background] ATS Committee on Proficiency Standards for Clinical Pulmonary Function Laboratories. ATS statement: guidelines for the six-minute walk test. Am J Respir Crit Care Med. 2002 Jul 1;166(1):111-7. doi: 10.1164/ajrccm.166.1.at1102. No abstract available. PMID 12091180
- [Background] Kazerooni EA, Martinez FJ, Flint A, Jamadar DA, Gross BH, Spizarny DL, Cascade PN, Whyte RI, Lynch JP 3rd, Toews G. Thin-section CT obtained at 10-mm increments versus limited three-level thin-section CT for idiopathic pulmonary fibrosis: correlation with pathologic scoring. AJR Am J Roentgenol. 1997 Oct;169(4):977-83. doi: 10.2214/ajr.169.4.9308447.
- [Background] Collard HR, Anstrom KJ, Schwarz MI, Zisman DA. Sildenafil improves walk distance in idiopathic pulmonary fibrosis. Chest. 2007 Mar;131(3):897-899. doi: 10.1378/chest.06-2101. PMID 17356110
- [Background] Madden BP, Allenby M, Loke TK, Sheth A. A potential role for sildenafil in the management of pulmonary hypertension in patients with parenchymal lung disease. Vascul Pharmacol. 2006 May;44(5):372-6. doi: 10.1016/j.vph.2006.01.013. Epub 2006 Mar 29. PMID 16574495
- [Background] Snyder EM, Olson TP, Johnson BD, Frantz RP. Influence of sildenafil on lung diffusion during exposure to acute hypoxia at rest and during exercise in healthy humans. Eur J Appl Physiol. 2008 Jul;103(4):421-30. doi: 10.1007/s00421-008-0735-5. PMID 18369657

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil: 20 mg of oral sildenafil, single dose at baseline
  Oral sildenafil 20 mg: A single dose of sildenafil will be given after recording baseline diffusion capacity and 6 minute walk. Measurements will be repeated one hour after the drug.
Period: Overall Study
Arm/Group | Sildenafil
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sildenafil
Number analyzed (Participants) | 15
Age, Continuous [Mean (Full Range); unit: years] | 58.6 [45.6 to 71.6]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 8

OUTCOME MEASURES:

1. Primary Outcome: Change in Diffusion Capacity Measured at Baseline and One Hour.
Description: Determine the acute effect of oral sildenafil on diffusion capacity in patients with diffuse parenchymal lung disease and concomitant pulmonary hypertension
Time Frame: Baseline and one hour
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Sildenafil
Number analyzed (Participants) | 15
ml/min/mmHg | -0.26 (0.94)
Statistical Analysis 1: Comparison: Sildenafil; Assuming 15% change in absolute value of DLCO representing a significant clinical difference and a standard deviation of 17.4% in normal nonsmoking individuals [Miller A, Thornton JC, Warshaw R, et al. Am Rev Respir Dis. 1983;127 (suppl 3):270-277.], 13 subjects needed to be studied to reject the null hypothesis when there is no significant difference between DLCO measurements before and after sildenafil, with power 0.8 and type I error probability 0.05 (SAS 9.2, SAS Institute Inc., Cary, NC); Test type: Superiority or Other; p = 0.30, t-test, 2 sided

2. Secondary Outcome: Change in 6 Minute Walk Distance
Description: The change in 6 minutes walk distance from baseline one hour after receiving 20 mg of sildenafil orally will be measured.
Time Frame: Baseline and one hour
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | Sildenafil
Number analyzed (Participants) | 15
feet
  Baseline | 1195 (407)
  One Hour | 1214 (383)
Statistical Analysis 1: Comparison: Sildenafil; The average 6 minute walk distance at baseline was 1195±407 feet. After oral administration of sildenafil, 6 minute walk distance was 1214±383 feet (p=0.63); Test type: Superiority or Other; p = 0.63, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Sildenafil
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No